CLINICAL TRIAL: NCT06064617
Title: Accommodative Behaviors in Multifocal Contact Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Ann Morrison, Assistant Professor, Ohio State University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 2023H0080
Record Dates: First submitted 2023-09-14; First posted 2023-10-03 (Actual); Results first posted 2026-01-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Accommodation Disorder

STUDY DESIGN:
Intervention Model Description: This study will be an observational single-center investigation using a cross sectional design and each subject will undergo two test sessions and will wear two different contact lenses. Each test session will take approximately 2 hours.
  The two arms are as follow:
  * Center-Distance (+2.50D add) then Center-Near (+2.50D add)
  * Center-Near (+2.50D add) then Center-Distance (+2.50D add)
Who Masked: Participant
Masking Description: Participants will not know what lens they are in
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Center Distance then Center Near Multifocal Contact Lens (Experimental): All participants will wear a Biofinity center distance multifocal contact lens with a +2.50 add and measurements will be obtained. Then participants will wear a Biofinity center near multifocal contact lens with a +2.50 add and measurements will be obtained.
  Interventions: Device: Center-Near (+2.50D) Coopervision Biofinity Multifocal Contact Lens; Device: Center Distance (+2.50 D) Coopervision Biofinity Multifocal Contact Lens
- Center Near then Center Distance Multifocal Contact Lens (Experimental): All participants will wear a Biofinity center near multifocal contact lens with a +2.50 add and measurements will be obtained. Then all participants will wear a Biofinity center distance multifocal contact lens with a +2.50 add and measurements will be obtained.
  Interventions: Device: Center-Near (+2.50D) Coopervision Biofinity Multifocal Contact Lens; Device: Center Distance (+2.50 D) Coopervision Biofinity Multifocal Contact Lens

INTERVENTIONS:
Device: Center-Near (+2.50D) Coopervision Biofinity Multifocal Contact Lens — Center-Near multifocal design
Device: Center Distance (+2.50 D) Coopervision Biofinity Multifocal Contact Lens — Center-Distance multifocal design

SUMMARY:
Addition lenses are often used to treat a range of eye conditions. Addition lenses are specifically used to help patients who do not have the ability to focus their eyes to see clearly up close. Eye focusing is called accommodation. Addition lenses are easy to prescribe in a pair of glasses and are often called the bifocal portion of the glasses. Addition lenses can be used for adults who have presbyopia (they cannot read up close without the aide of a bifocal) and for patients of all ages who have eye focusing problems (e.g. accommodative insufficiency, accommodative infacility, accommodative dysfunction).

Addition powers can also be put into contact lenses. Contact lenses that have addition powers in them are called multifocal contact lenses. These are often marketed for patients that are 40 and over who have presbyopia, and are prescribed to help patients see up close as well as far away in their contact lenses. Multifocal contact lenses are also used in children with nearsightedness because studies have shown that some multifocal designs can slow down the progression of nearsightedness. As stated before, addition lenses can be used to treat eye focusing problems in patients of all ages, before presbyopia. What is unclear is whether the addition power in contact lenses has the same treatment effect as an addition power in a pair of glasses when they are being used to treat eye focusing problems. This study will assess how different kinds of multifocal contact lenses (center distance or center near) will change eye focusing and eye teaming in young adult patients.

DETAILED DESCRIPTION:
Soft multifocal contact lenses are used for a variety of reasons in patient care. In fact, studies have shown that soft multifocal contact lenses alter accommodation. While most often used to correct presbyopic vision, these lenses are also used in the management of accommodative and binocular vision disorders along with myopia management. Multifocal contact lenses correct vision at different distances by introducing a power gradient over the eye thus providing a range of clear vision at both distance and near.

For center near designs, the near addition is placed in the center of the lens, and the power becomes more negative in the periphery. Generally, it is thought that center near designs provide the most accommodative relief and superior near vision because the near addition is centered in the pupil. These lenses allow maximum near correction, even with miotic pupil size changes associated with accommodation. Conversely, for center distance designs, the distance prescription is placed in the center, and the power of the lens becomes more positive in the periphery to provide the near addition. To date, most studies have used center-distance lens designs to evaluate accommodative ability and function. Accommodative function while wearing center near lenses has likely not been studied often because these lens designs are used most in populations with no or waning accommodative ability (i.e. presbyopic patients). In this population lenses are used, specifically, to account for that accommodative inability.

Center near and distance designs have varying advantages and disadvantages for presbyopic vision correction. Selection of lens design can be based on a patient's individual visual needs. There is conflicting evidence on whether the add power in soft multifocal contact lenses can be used to manage accommodative and binocular vision disorders. These lenses do offer relief of accommodative demand associated with both accommodative and binocular vision disorders. It has been hypothesized that center near multifocal contact lenses provide a greater therapeutic effect as the central portion of the lens is the addition power. There have been case reports demonstrating benefits of multifocal contact lenses in accommodative insufficiency and convergence excess. Center distance lenses are used most often for myopia management. In these situations, the interest has been to determine if the child can maintain normal accommodative function while wearing the lenses. This study will aim to determine how accommodative function varies with center distance and center near multifocal contact lenses.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18 to ≤ 30 years old
* Acuity of 20/25 or better in both eyes with habitual contact lens prescription
* No history of ocular disease or active ocular inflammation
* No history of ocular or refractive surgery
* No current history of rigid contact lens wear
* Astigmatism ≤1.00 D
* Free of binocular vision disorder (strabismus, amblyopia, vergence dysfunction, accommodative dysfunction)

Exclusion Criteria:

* No prior or concurrent participation in myopia control or use of low dose atropine, multifocal contact lenses
* No use of any medications suspected to affect accommodation

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ann M Morrison, OD, PhD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided
If there is a benefit to sharing data, then data can be shared after publication of the primary outcome paper.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Potential participants will be recruited in the following manners:
  * Word of mouth by the investigators among employees and visitors to the College of Optometry
  * Flyers
  * Email announcements distributed to the faculty, staff, and students at OSU
  * Electronic advertisement in the OSU Healthbeat
  * Phone calls to potentially eligible participants who are identified from a review of clinical records at the College of Optometry to identify those who wear soft contact lenses.
Pre-assignment Details: All participants had a baseline examination where baseline clinical measures were taken. At the follow up appointment, they would wear center-distance and center-near lenses in which measurements from the baseline exam were repeated. The order of the wear lenses (center-distance and center-near) were randomized between subjects.
Groups:
- Center Distance, Then Center Near: Participants had clinical measurements taken with Center Distance lenses, then Center Near Lenses
- Center Near, Then Center Distance: Participants had clinical measurements taken with Center Distance lenses, then Center Near Lenses all within a visit that was 2 hours or less.
Period: First Intervention (1 hour)
Arm/Group | Center Distance, Then Center Near | Center Near, Then Center Distance
Started | 11 | 9
Completed | 11 | 9
Not Completed | 0 | 0
Period: Second Intervention (1 hour)
Arm/Group | Center Distance, Then Center Near | Center Near, Then Center Distance
Started | 11 | 9
Completed | 11 | 9
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: 20 Participants were measured in all three treatments (single vision, center-distance, and center-near)
Groups:
- Center Near, Then Center Distance: Participants had clinical measurements taken with Center-Near lenses, Then Center Distance lenses
- Total: Total of all reporting groups
Arm/Group | Center Distance, Then Center Near | Center Near, Then Center Distance | Total
Number analyzed (Participants) | 11 | 9 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 24.1 (1.4) | 23.2 (0.4) | 23.7 (1.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 5 | 13
  Male | 3 | 4 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 11 | 9 | 20
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 0 | 2
  White | 7 | 9 | 16
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Objective Accommodative Response (in Diopters) on the Grand Seiko Autorefractor at 2.5 Diopters (40 cm)
Description: Accommodative function will be compared using the Grand Seiko Autorefractor between the center distance and center near group. The instrument will record the patient's refractive error at near (40 cm), which is commonly used for near assessment in clinic. Patients place their head on a chin rest and look at targets at different distances. The examiner then pushes a button and the refractive error (in Diopters) is recorded from the instrument and placed in an excel file to be analyzed.
Time Frame: Up to two hours (1 hour in each lens)
Population: Every participant wore the center distance and center near lenses, we are comparing the clinical measures in all participants wearing the distance lenses to the clinical measures in all participants wearing the center near lenses.
Measure: Mean (Standard Deviation); unit: Diopters
Groups:
- Center Distatnce: Participants had clinical measurements taken with Center Distance lenses
- Center Near: Participants had clinical measurements taken with Center-Near lenses
Arm/Group | Center Distatnce | Center Near
Number analyzed (Participants) | 20 | 20
Diopters | 1.20 (0.17) | 1.03 (0.12)

2. Secondary Outcome: Accommodation (in Diopters) Measured by Monocular Estimation Method (MEM)
Description: Accommodation was assessed by monocular estimation method which is done with a clinical retinoscope, in which the examiner looks at the light reflex of the retina and the patient reads small print at 40 centimeters and the examiner uses lenses to neutralize the reflex
Time Frame: Up to two hours
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Diopters
Groups:
- Center Distance: Participants had clinical measurements taken with Center Distance lenses
Arm/Group | Center Distance | Center Near
Number analyzed (Participants) | 20 | 20
Diopters | 0.59 (0.08) | 0.18 (0.08)

3. Secondary Outcome: Accommodation (in Diopters) Measured by Monocular Push-Up
Description: Accommodation measured with a monocular push-up was measured by the examiner bringing a small target close to the eye and the patient reports when the target gets blurry. These eye focusing tests and outcomes will be compared in the lens types.
Time Frame: Up to 2 hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Diopters
Arm/Group | Center Distance | Center Near
Number analyzed (Participants) | 20 | 20
Diopters | 12.26 (0.45) | 10.95 (0.45)

4. Secondary Outcome: Accommodation (in Cycles Per Minute) Measured by Accommodative Facility
Description: Accommodation was assessed by accommodative facility which uses lenses to determine how many times a patient can clear a target in one minute by having the patient look at print 40 centimeters away and the examiner places a plus lens in front of the eye and the patient reports when the text is clear and the examiner flips the lens to a minus lens and the patient reports when the text is clear and this is done for one minute and cycles per minute are recorded
Time Frame: Up to 2 hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Cycles per Minute
Arm/Group | Center Distance | Center Near
Number analyzed (Participants) | 20 | 20
Cycles per Minute | 14.05 (0.78) | 12.15 (0.78)

5. Secondary Outcome: Phoria (in Prism Diopters) Measured by Modified Thorington at Distance
Description: Vergence measures will be completed by Modified Thorington will be assessed at distance (20 feet) which is a card with a light in the center. The patient holds up a red lens over their eye and they report where they see the line crossing the cards. This is recorded in prism diopters. This is tested with all lens types.
Time Frame: Up to 2 Hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Prism Diopters
Arm/Group | Center Distance | Center Near
Number analyzed (Participants) | 20 | 20
Prism Diopters | 0.53 (0.25) | 0.23 (0.25)

6. Secondary Outcome: Phoria (in Prism Diopters) Measured by Modified Thorington at Near
Description: Vergence measures was completed with Modified Thorington will be assessed at near (40 centimeters), which is a card with a light in the center. The patient holds up a red lens over their eye and they report where they see the line crossing the cards. This is recorded in prism diopters. This is tested with all lens types.
Time Frame: Up to 2 hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Prism Diopters
Arm/Group | Center Distance | Center Near
Number analyzed (Participants) | 20 | 20
Prism Diopters | -1.25 (0.88) | 0.05 (0.88)

ADVERSE EVENTS:
Time Frame: Enrollment to end of follow up. Each participant was seen for 2 visits, on two separate days. Each visit was no longer than 2 hours or 120 minutes each, so participants were seen for no more than 4 hours for the entire study. No participants' visits were separated by more than 2 weeks.
Description: Adverse Events were described the same as Clinical Trials.gov has listed.
  Adverse Events are typically reported "per intervention" but in order to ensure that there was no double counting of participants, the arms were listed (as advised by clinicaltrials.gov) to show the order of which treatment was received (because ALL participants received all the treatments and order was randomized). But all participants are accounted for in the reporting, as well as adverse events.
Arm/Group | Center Distance | Center Near
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20

LIMITATIONS AND CAVEATS:
The participants were not allowed to adapt to the contact lenses outside of the office - all testing was done in office and participants were not allowed to take the contact lenses out of the office.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-11-30): https://cdn.clinicaltrials.gov/large-docs/17/NCT06064617/Prot_SAP_001.pdf